CLINICAL TRIAL: NCT03585270
Title: A Prospective, Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Phase 3 Study to Assess the Efficacy and Safety of Clazosentan in Preventing Clinical Deterioration Due to Delayed Cerebral Ischemia (DCI), in Adult Subjects With Aneurysmal Subarachnoid Hemorrhage (aSAH)
Brief Title: Clinical Research Study With Clazosentan to Evaluate Its Effects on Preventing Complications Due to the Narrowing of the Blood Vessels (Vasospasm) in the Brain, Caused by Bleeding Onto the Surface of the Brain
Acronym: REACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ID-054-304; 2018-000241-39 (EudraCT Number)
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — clazosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be performed in a double-blind fashion. The investigator, study personnel, subjects, clinical research associates (CRAs), sponsor personnel, and vendor / Contract Research Organization (CRO) personnel involved in the conduct of the study will remain blinded to the study treatment received by the subjects during the double-blind treatment period until study closure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clazosentan (Experimental): Participants will receive clazosentan for up to 14 days, followed by a safety follow-up period of 24 hours, and an extended follow-up period to the end-of-study visit at Week 24 post aneurysmal subarachnoid hemorrhage (aSAH).
  Interventions: Drug: Clazosentan
- Placebo (Placebo Comparator): Participants will receive clazosentan matching-placebo for up to 14 days, followed by a safety follow-up period of 24 hours, and an extended follow-up period to the end-of-study visit at Week 24 post aneurysmal subarachnoid hemorrhage (aSAH).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clazosentan — Clazosentan will be administered as a continuous intravenous infusion at the dose of 15 mg/hour for up to 14 days.
  Other Names: ACT-108475
  Arms: Clazosentan
Drug: Placebo — Placebo will be administered at the same infusion rate as clazosentan for up to 14 days.
  Arms: Placebo

SUMMARY:
This study will evaluate if clazosentan (on top of normal routine medical care) can reduce the risk of developing complications related to cerebral vasospasm and permanent brain damage as compared to normal routine medical care alone.

DETAILED DESCRIPTION:
When a blood vessel just outside the brain bursts and causes bleeding onto its surface, the space surrounding the brain (the subarachnoid space) fills with blood. This condition is called subarachnoid hemorrhage. The bleeding due to the rupture of a pouch-like structure or a bulge (called an aneurysm) that formed on one of the blood vessels is condition called aneurysmal subarachnoid hemorrhage (aSAH).

In this study, clazosentan is being tested against normal routine medical care to determine if clazosentan can reduce the risk of developing complications related to vasospasm and permanent brain damage.

Participation will last for approximately 6 months from the episode of bleeding. For subjects randomized in the high-risk prevention group, treatment will start within 96 hours following the time of the aneurysm rupture, and be administered where possible, for 14 days. For subjects randomized in the early treatment group, treatment must begin within 24 hours of the time of the angiogram documenting the cerebral vasospasm necessary for entry into the study. Treatment will be administered for a minimum of 6 days and a maximum of 14 days. Recruitment in the early treatment group has been discontinued.

The end-of-study will be conducted as a telephone interview 6 months after the episode of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study must be obtained from the subject or proxy/legal representative at any time from hospital admission to prior to initiation of any study-mandated procedure,
* Males and females aged 18 to 70 years (inclusive, at hospital admission),
* Participants with a ruptured saccular aneurysm, angiographically confirmed by DSA or CTA, which has been successfully secured within 72 hours of rupture, by surgical clipping or endovascular coiling,
* WFNS (World Federation of Neurosurgical Societies) grades 1-4 (based on Glasgow Coma Scale [GCS]) assessed after recovery from the aneurysm-securing procedure and after external ventricular drainage for hydrocephalus, if required.
* Participants must meet the criteria for the high-risk prevention group: Subjects with a "thick and diffuse clot" (thick and diffuse is defined as a thick confluent clot, more than 4 mm in thickness, involving 3 or more basal cisterns) on the hospital admission CT scan, absence of cerebral vasospasm at the time of randomization, and possibility to start study drug in the ICU (or equivalent environment where all protocol assessments can be performed and the Patient Management Guidelines followed), within 96 hours after the time of the aneurysm rupture.
* The recruitment into the early treatment group, i.e. participants without a thick and diffuse clot on the hospital admission CT scan who develop asymptomatic or minimally symptomatic moderate to severe angiographic vasospasm, within the 14-day period post-aneurysm rupture, and for whom it is possible to start study drug in the ICU (or equivalent environment where all protocol assessments can be performed and the Patient Management Guidelines followed), within 24 hours of this angiographic diagnosis, has been discontinued.
* Presence of a cerebral CT scan performed at least 8 hours post aneurysm securing procedure and within 24 hours prior to randomization.
* Absence of a significant (e.g., symptomatic or large) new or worsened cerebral infarct or re-bleeding of the repaired aneurysm on the post-procedure CT scan.
* A woman of childbearing potential is eligible only if the pregnancy test performed during the screening period is negative. Agreement must be obtained to take the necessary precautions to avoid pregnancy from hospital discharge until 30 days post-study drug discontinuation. If breastfeeding, agreement must be obtained to refrain for the duration of the treatment with study drug and until 30 days post-study drug discontinuation.
* Males are eligible for study participation only if they agree to take the necessary precautions to avoid pregnancy in a female partner from hospital discharge until 30 days post-study drug discontinuation.

Exclusion Criteria:

* Aneurysmal subarachnoid hemorrhage (aSAH), aneurysm-securing procedure, vasospasm:

  * Participants with SAH due to causes other than a saccular aneurysm (e.g., trauma or rupture of fusiform or mycotic aneurysms, SAH associated with arterio-venous malformation, vertebral dissections),
  * Significant bleeding post aneurysm-securing procedure (e.g., due to intra-ventricular drain, intra-cerebral hemorrhage, epidural hematoma, vessel dissection or rupture, re-bleeding of the repaired aneurysm), based on investigator judgment,
  * Intra-or peri-aneurysm securing procedure complication requiring non-routine medical or interventional treatment such as administration of an antithrombotic or anti-platelet agent (e.g., abciximab), which is not completely resolved prior to randomization,
  * Intraventricular hemorrhage on the hospital admission CT scan, filling more than 50% of both lateral ventricles and with involvement of the 3rd and 4th ventricles.
  * Intracerebral hemorrhage on the hospital admission CT scan, with an approximate volume of > 50 mL,
  * Presence of cerebral vasospasm at hospital admission (initial admission or transfer from another hospital) believed to be associated with a prior bleed (i.e., occurring before the bleed for which the subject is currently hospitalized). Vasospasm occurring during the aneurysm securing procedure is not an exclusion criterion,
* Neurological and functional status:

  * Participants with a new major neurological deficit occurring post aneurysm-securing procedure which is attributable to the procedure and does not improve to pre-procedure status before randomization,
  * Participants with a GCS score of ≤ 9 at the time of randomization and without intracranial pressure (ICP) monitoring,
  * Modified Rankin Score of 3 or higher, prior to the aSAH (i.e., due to a chronic condition),
* Other clinical considerations:

  * Participants with total bilirubin > 2 times the upper limit of normal, and/or a known diagnosis or clinical suspicion of liver cirrhosis or moderate to severe hepatic impairment,
  * Hypotension (systolic blood pressure [SBP] ≤ 90 mmHg) at time of randomization that is refractory to treatment,
  * Unresolved pulmonary edema or significant pneumonia still present at the time of randomization, or severe hypoxia at the time of randomization in intubated subjects, defined as PaO2/FiO2 ≤ 200,
  * High sustained ICP (> 25 mmHg lasting > 20 minutes) at time of randomization, despite optimal treatment, in subjects with ICP monitoring,
  * Severe cardiac failure requiring inotropic support at the time of random

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2019-02-03 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (80):
- United States (16):
  - Stanford Hospital & Clinics - Stanford School of Medicine Dept. of Neurosurgery, Stanford, California
  - Mayo clinic, Dept of Neurosurgery, Jacksonville, Florida
  - University of Illinois - Department of Neurosurgery, Chicago, Illinois
  - University of Maryland Medical Systems - Neurosurgery, Baltimore, Maryland
  - Boston University School of Medicine / Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center Dept of Neurosurgery, Boston, Massachusetts
  - Northwell Health, Department of Neurosurgery, Manhasset, New York
  - Mt Sinai Hospital, New York, New York
  - Columbia University Medical Center Dept. of Neurology - Neurological Intensive Care Unit, New York, New York
  - University Hospitals Case Medical Center - Department of Neurosurgery, Cleveland, Ohio
  - The Ohio State University - Wexner Medical Center, Columbus, Ohio
  - Oklahoma University Health Sciences Center - Department of Neurology, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Neurosurgery, Hershey, Pennsylvania
  - Vanderbilt University Medical Center - Department of Neurosurgery, Nashville, Tennessee
  - Virginia Commonwealth University, Department of Neurosurgery, Richmond, Virginia
- Austria (2):
  - Medizinische Universität Innsbruck; Universitätsklinik für Neurologie und Psychiatrie, Innsbruck
  - Kepler Universitätsklinikum, Universitätsklinik für Neurochirurgie, Linz
- Belgium (4):
  - Hospital Erasme, Service de Soins Intensifs, Brussels
  - Hospital - Cliniques Universitaires Saint-Luc, Service de Neurochirurgie, Brussels
  - Neurology Department, University Hospital, Ghent
  - University Hospital Sart Tilman Liege, Liège
- Canada (4):
  - University of Alberta Hospital Department of Neurological Surgery, Edmonton, Alberta
  - Winnipeg Regional Health Authority Health Sciences Centre, Winnipeg, Manitoba
  - Halifax Infirmary, Nova Scotia Health Authority, Halifax, Nova Scotia
  - Royal University Hospital Department of Neurology, Saskatoon, Saskatchewan
- Czechia (5):
  - Fakultní nemocnice Brno Neurochirurgická klinika, Brno
  - Fakultní nemocnice Ostrava Neurochirurgická klinika, Ostrava-Poruba
  - University Hospital in Pilsen, Department of Neurosurgery, Pilsen
  - Ústřední vojenská nemocnice Praha Neurochirurgická klinika, Prague
  - Masarykova nemocnice v Ústí nad Labem Neurochirurgie, Ústí nad Labem
- Odense Universitets Hospital Neurokirurgisk afdelning, Odense, Denmark
- Finland (4):
  - Helsingin yliopistollinen keskussairaala Neurokirurgian klinikka, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampereen yliopistollinen sairaala Neurokirurgian klinika, Tampere
  - Turku University Hospital Neurosurgery, T-hospital, Turku
- France (7):
  - Hôpital neurologique Pierre Wertheimer Service de Reanimation, Bron
  - Hôpital Gabriel Montpied, ICU DEPT, Neuro reanimation departement, Clermont-Ferrand
  - Hôpital de la Timone 2, Intensive Care Unit SAR 1, Marseille
  - Hôpital Nord Laennec - CHU de Nantes, Nantes
  - Hospital Lariboisiere Paris, Paris
  - Hôpital Pitié-Salpêtrière, Service de neuroréanimation chirurgicale Babinski, Paris
  - Univ Hosp Toulouse, University Hospital Purpan Pierre Paul Riquet Hospital, Toulouse
- Germany (13):
  - Klinik für Diagnostische Radiologie und Neuroradiologie, Augsburg, Augsburg
  - Charite Universitätsmedizin Berlin - Klinik und Poliklinik für Neurochirurgie, Berlin
  - Heinrich-Heine Universität Düsseldorf -Klinik für Neurochirugie, Düsseldorf
  - University of Erlangen-Nürnberg, Dpt. of Neurosurgery, Erlangen
  - University Hospital of Essen, Department of Neurosurgery, Essen
  - Universitätsklinik Frankfurt, Klinik und Poliklinik für Neurochirurgie, Dept of neurosurgery, Frankfurt
  - Bezirkskrankenhaus Günzburg - Klinik für Neurochirugie, Günzburg
  - Asklepios Klinik St. Georg - Neurochirugie, Hamburg
  - University Hospital of Hamburg-Eppendorf, Dpt. of Neurosurgery, Hamburg
  - Neurochirurgische Universitätklinik des Heidelberg, Dept of Neurosurgery, Heidelberg
  - Universitätsklinikum Schleswig Hollstein Lübeck (UKSH) Klinik für Neurochirugie, Lübeck
  - University Regensburg, Dpt. of Neurosurgery, Regensburg
  - Universitätsklinikum Rostock, Abteilung für Neurochirurgie, Rostock
- Hungary (2):
  - Debreceni Egyetem, Idegsebészet, Debrecen
  - Pécsi Tudományegyetem Klinikai Központ, Idegsebészeti Klinika, Pécs
- Israel (4):
  - Rambam Healthcare Campus, Neurology Department, Haifa
  - Hadassah Medical Center, Jerusalem
  - Beilinson Hospital, Rabin Medical Center, Department of Neurosurgery, Petah Tikva
  - The Chaim Sheba Medical Centre - Neurosurgery, Ramat Gan
- Italy (4):
  - ASST Monza, Hospital San Gerardo, TERAPIA INTENSIVA Neurochirurgica, Monza
  - Azienda Ospedaliera Padova-Università degli Studi di Padova - Istituto di Anestesia e Rianimazione, Padua
  - Azienda Ospedaliero Universitaria di Parma, struttura complessa Neurochirurgia, Parma
  - Fondazione Policlinico Universitario Agostino Gemelli Università Cattolica del Sacro Cuore, UOS Terapia Intensiva Neurochirurgic, Rome
- Poland (3):
  - Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego, Lodz
  - Oddział Neurochirurgii i Neurotraumatologii z Pododdziałem Leczenia Chorób Naczyniowych Centralnego Układu Nerwowego, Poznan
  - Katedra i Klinika Neurochirurgii Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Warsaw
- Spain (8):
  - Hospital Universitario Germans Trias i Pujol - Neurology Department, Badalona
  - Hospital Vall d'Hebron Departamento Neuroradiología, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - University Hospital of Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario 12 de Octubre, Departamento Neurosurgery Division Neuroradiology, Madrid
  - Hospital Universitari son Espases, Palma de Mallorca
  - Corporació Sanitària Parc Taulí, Hospital Parc Taulí, Sabadell
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Verksamheten för neurokirurgi, Neurosjukvården, Gothenburg
  - Linköping Universitetssjukhuset, Neurokirurgiska kliniken, Linköping
  - Lunds Universitetssjukhus, Neurokirurgiska avd. NIVA, Lund

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayer SA, Bruder N, Citerio G, Defreyne L, Dubois C, Gupta R, Higashida R, Marr A, Nguyen TN, Roux S, Smrcka M, Torne RT, Aldrich EF; on behalf of the REACT investigators. REACT: a randomized trial to assess the efficacy and safety of clazosentan for preventing clinical deterioration due to delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage. J Neurosurg. 2024 Aug 9;142(1):98-109. doi: 10.3171/2024.4.JNS232191. Print 2025 Jan 1. PMID 39126720
- [Derived] Bruder N, Higashida R, Santin-Janin H, Dubois C, Aldrich EF, Marr A, Roux S, Mayer SA. The REACT study: design of a randomized phase 3 trial to assess the efficacy and safety of clazosentan for preventing deterioration due to delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage. BMC Neurol. 2022 Dec 20;22(1):492. doi: 10.1186/s12883-022-03002-8. PMID 36539711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 03 February 2019 to 18 November 2022.
Pre-assignment Details: Of 453 participants screened, 409 were enrolled in the study and randomized to study treatment.
Groups:
- Clazosentan: All participants from the randomized analysis set who started clazosentan 15 mg per hour infusion for up to 14 days.
- Placebo: All participants from the randomized analysis set who started matching placebo infusion for up to 14 days.
Period: Overall Study
Arm/Group | Clazosentan | Placebo
Started (Randomized Analysis Set) | 203 | 206
Not Treated (Participants were randomized but not treated) | 1 | 2
Started Treatment (Assigned Treatment Groups) (Full Analysis Set: all randomized participants who started study treatment, evaluated according to assigned treatment.) | 202 | 204
Started Treatment (Actual Treatment Received) (Safety Analysis Set: all randomized participants who started study treatment, evaluated according to the actual treatment received. Note that 5 participants randomized to placebo received at least 1 infusion of clazosentan and were analyzed as part of the clazosentan arm for this analysis set.) | 207 | 199
Completed | 187 | 189
Not Completed | 16 | 17
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Withdrawal by proxy/legal representative | 1 | 0
Not completed — Adverse Event | 5 | 2
Not completed — Lost to Follow-up | 1 | 4
Not completed — Death | 5 | 3
Not completed — Other reasons | 2 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Clazosentan | Placebo | Total
Number analyzed (Participants) | 202 | 204 | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (10.4) | 53.7 (10.0) | 53.3 (10.2)
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 64 years | 171 | 175 | 346
  Between 65 to 84 years | 31 | 29 | 60
  85 years and older | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 137 | 275
  Male | 64 | 67 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 23 | 48
  Not Hispanic or Latino | 155 | 159 | 314
  Unknown or Not Reported | 22 | 22 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 176 | 169 | 345
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 21 | 37
Region of Enrollment [Number; unit: participants]
  Austria | 6 | 6 | 12
  Belgium | 15 | 17 | 32
  Canada | 8 | 12 | 20
  Czechia | 23 | 24 | 47
  Denmark | 2 | 3 | 5
  Finland | 14 | 11 | 25
  France | 15 | 18 | 33
  Germany | 26 | 16 | 42
  Hungary | 4 | 3 | 7
  Israel | 6 | 7 | 13
  Italy | 11 | 18 | 29
  Poland | 5 | 11 | 16
  Spain | 24 | 24 | 48
  Sweden | 8 | 10 | 18
  United States | 35 | 24 | 59
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] — at hospital admission Population: Data not available for 6 participants
  kilograms per square meter
    number analyzed (Participants) | 200 | 200 | 400
    (all) | 26.8 (5.7) | 26.8 (5.6) | 26.8 (5.6)
Total Glasgow Coma Scale (GCS) Score [Mean (Standard Deviation); unit: units on a scale] — The GCS was performed at hospital admission. The GCS was used to measure the level of consciousness. Scores range from 3 (worst score) to 15 (best score). Population: Data not available for 2 participants.
  units on a scale
    number analyzed (Participants) | 201 | 203 | 404
    (all) | 13.4 (3.0) | 13.1 (3.3) | 13.2 (3.2)
World Federation of Neurological Societies (WFNS) Grade [Count of Participants; unit: Participants] — The WFNS grade was assessed by the investigator at hospital admission. The WFNS grade ranges from I (best) to V (worst).
  Participants
    Grade I and II | 161 | 158 | 319
    Grade III to V | 41 | 46 | 87
Aneurysmal subarachnoid hemorrhage diagnosed subgroups [Count of Participants; unit: Participants] — High-risk prevention participants were diagnosed at an early stage of the disease continuum and were those who were at a high risk of developing cerebral vasospasm. These participants were characterized by the presence of a large quantity of subarachnoid blood on their hospital admission Computed Tomography (CT) scan (with a "thick and diffuse clot" defined as a thick confluent clot, more than 4 mm in thickness and involving more than 3 or more basal cisterns).
  The confirmed vasospasm participants did not have a "thick and diffuse clot" on their hospital admission CT scan.
  Participants
    Confirmed vasospasm group | 6 | 5 | 11
    High risk of vasospasm (high-risk prevention) group | 196 | 199 | 395

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Clinical Deterioration Due to Delayed Cerebral Ischemia (DCI) From Study Drug Initiation up to 14 Days Post-study Drug Initiation
Description: Clinical deterioration due to delayed cerebral ischemia is defined as a worsening of at least 2 points compared to the reference score, on the modified Glasgow Coma Scale or the abbreviated National Institutes of Health Stroke Scale (aNIHSS), lasting for at least 2 hours, which cannot be entirely attributed to causes other than cerebral vasospasm. It is centrally adjudicated by the Clinical Event Committee (CEC) based on a written charter and review of clinical data, case narratives, angiograms and Computed Tomography scans.
Time Frame: Up to 14 days post-study drug initiation
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Clazosentan | Placebo
Number analyzed (Participants) | 202 | 204
Participants | 32 | 35
Statistical Analysis 1: Comparison: Clazosentan vs Placebo; Test type: Superiority; p = 0.7338, Cochran-Mantel-Haenszel; Relative Risk Reduction = 0.072, 95% CI 2-sided [-0.426 to 0.396] — Homogeneity of the treatment effect across strata was investigated using the Breslow-Day test (p-value = 0.2785)

2. Secondary Outcome: Occurrence of Clinically Relevant Cerebral Infarction at Day 16 Post-study Drug Initiation
Description: A clinical relevant cerebral infarction was defined as: all-cause cerebral infraction greater than or equal to 5 cm^3 or cerebral infarction less than 5 cm^3 in participants with clinical deterioration due to delayed cerebral ischemia.
  Cerebral infarction refers to new or worsened infarcts and was determined by a central radiology review comparing the total volume of infarcts on the computed tomography (CT) scan performed 16 days after study drug initiation with the total volume on the CT scan performed just prior to randomization.
Time Frame: At Day 16 post study drug initiation
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Clazosentan | Placebo
Number analyzed (Participants) | 202 | 204
Participants | 15 | 23
Statistical Analysis 1: Comparison: Clazosentan vs Placebo; Test type: Superiority; p = 0.177, Cochran-Mantel-Haenszel; Relative Risk Reduction = 0.341, 95% CI 2-sided [-0.213 to 0.642] — Homogeneity of the treatment effect across strata was investigated using the Breslow-Day test (p-value = 0.8644)

3. Secondary Outcome: Long-term Clinical Outcome Assessed by the Modified Rankin Scale (mRS) at Week 12 Post-aneurysmal Subarachnoid Hemorrhage (aSAH)
Description: The modified Rankin Scale (mRS) was used to measure the degree of disability in participants who had a ruptured saccular aneurysm and were at a high risk of developing a delayed cerebral infarction (DCI). The mRS is scored by the physician. The mRS scores ranged from 0 (no symptoms) to 6 (dead). The mRS score was dichotomized into poor outcome (score greater and equal to 3) and good outcome (score less than 3).
Time Frame: At Week 12 post-aneurysmal subarachnoid hemorrhage (aSAH)
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Clazosentan | Placebo
Number analyzed (Participants) | 202 | 204
Participants
  Participants with a mRS score of equal and greater than 3 | 50 | 41
  Participants with a mRS score of less than 3 | 152 | 163
Statistical Analysis 1: Comparison: Clazosentan vs Placebo; Test type: Superiority; p = 0.1983, Cochran-Mantel-Haenszel; Relative Risk Reduction = -0.254, 95% CI 2-sided [-0.760 to 0.107] — Homogeneity of the treatment effect across strata was investigated using the Breslow-Day test (p-value = 0.8844)

4. Secondary Outcome: Long-term Clinical Outcome Assessed by the Glasgow Outcome Scale Extended (GOSE) at Week 12 Post-aSAH
Description: The Glasgow Outcome Scale - Extended (GOSE) is a scale scored by the physician. The GOSE scores range from 1 (dead) to 8 (upper good recovery).
  The long-term clinical outcome assessed by the GOSE was dichotomized into poor outcome (score ≤ 4) and good outcome (score > 4)
Time Frame: At Week 12 post-aneurysmal subarachnoid hemorrhage (aSAH)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Clazosentan | Placebo
Number analyzed (Participants) | 202 | 204
Participants
  Participants with a GOSE score less than and equal to 4 | 50 | 41
  Participant with a GOSE score greater than 4 | 152 | 163
Statistical Analysis 1: Comparison: Clazosentan vs Placebo; Test type: Superiority; p = 0.1983, Cochran-Mantel-Haenszel; Relative Risk Reduction = -0.254, 95% CI 2-sided [-0.760 to 0.107] — Homogeneity of the treatment effect across strata was investigated using the Breslow-Day test (p-value = 0.8844)

5. Other Pre Specified Outcome: Occurrence of Clinical Deterioration Due to Delayed Cerebral Ischemia (DCI) From Study Drug Initiation up to 14 Days Post-study Drug Initiation (Safety Analysis Set)
Description: Clinical deterioration due to delayed cerebral ischemia is defined as a worsening of at least 2 points compared to the reference score, on the modified Glasgow Coma Scale or the abbreviated National Institutes of Health Stroke Scale (aNIHSS), lasting for at least 2 hours, which cannot be entirely attributed to causes other than cerebral vasospasm. It is centrally adjudicated by the Clinical Event Committee (CEC) based on a written charter and review of clinical data, case narratives, angiograms and computed tomography (CT) scans.
Time Frame: Up to 14 days post-study drug initiation
Population: Safety Analysis Set: all randomized participants who started study treatment, evaluated according to the actual treatment received. Note that 5 participants randomized to placebo received at least 1 infusion of clazosentan and were analyzed as part of the clazosentan arm for this analysis set.
Measure: Count of Participants; unit: Participants
Groups:
- Clazosentan: Participants that received at least one clazosentan 15 mg per hour infusion.
- Placebo: Participants that received placebo infusions for up to 14 days.
Arm/Group | Clazosentan | Placebo
Number analyzed (Participants) | 207 | 199
Participants | 32 | 35
Statistical Analysis 1: Comparison: Clazosentan vs Placebo; Test type: Superiority; p = 0.5591, Cochran-Mantel-Haenszel; Relative Risk Reduction = 0.119, 95% CI 2-sided [-0.349 to 0.425] — Homogeneity of the treatment effect across strata was investigated using the Breslow-Day test (p-value = 0.1706)

6. Other Pre Specified Outcome: Occurrence of Clinical Deterioration Due to Delayed Cerebral Ischemia (DCI) From Study Drug Initiation up to 14 Days Post-study Drug Initiation Including Rescue Therapy for Non-relevant Vasospasm
Description: Clinical deterioration due to delayed cerebral ischemia is defined as a worsening of at least 2 points compared to the reference score, on the modified Glasgow Coma Scale or the abbreviated National Institutes of Health Stroke Scale (aNIHSS), lasting for at least 2 hours, which cannot be entirely attributed to causes other than cerebral vasospasm. It is centrally adjudicated by the Clinical Event Committee (CEC) based on a written charter and review of clinical data, case narratives, angiograms and Computed Tomograph (CT) scans.
Time Frame: Up to 14 days post-study drug initiation
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Clazosentan | Placebo
Number analyzed (Participants) | 202 | 204
Participants | 34 | 47
Statistical Analysis 1: Comparison: Clazosentan vs Placebo; Test type: Superiority; p = 0.1179, Cochran-Mantel-Haenszel; Relative Risk Reduction = 0.267, 95% CI 2-sided [-0.085 to 0.505] — Homogeneity of the treatment effect across strata was investigated using the Breslow-Day test (p-value = 0.4580)

7. Other Pre Specified Outcome: Occurrence of Clinical Deterioration Due to Delayed Cerebral Ischemia (DCI) From Study Drug Initiation up to 14 Days Post-study Drug Initiation Based on Neurological Scales and Death
Description: as for outcome 6
Time Frame: Up to 14 days post-study drug initiation
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Clazosentan | Placebo
Number analyzed (Participants) | 202 | 204
Participants | 28 | 33
Statistical Analysis 1: Comparison: Clazosentan vs Placebo; Test type: Superiority; p = 0.5217, Cochran-Mantel-Haenszel; Relative Risk Reduction = 0.139, 95% CI 2-sided [-0.365 to 0.457] — Homogeneity of the treatment effect across strata was investigated using the Breslow-Day test (p-value = 0.1685)

ADVERSE EVENTS:
Time Frame: Adverse events were considered treatment-emergent, if the onset date was from the start of the first infusion on Day 1 to up to 24 hours after study treatment discontinuation. Study treatment was planned for up to 14 days.
Description: Safety Analysis Set: evaluated according to the actual treatment received. Note that 5 participants randomized to placebo received at least 1 infusion of clazosentan and were analyzed as part of the clazosentan arm for this analysis set.
  All-cause mortality: 10 participants died (7 clazosentan, 3 placebo). For 2 of the participants in the clazosentan group, the reason for study discontinuation was reported as Adverse event, i.e., with fatal outcome (see Participant flow).
Groups:
- Clazosentan: Participants that received at least one dose of clazosentan.
- Placebo: Participants that received placebo.
Arm/Group | Clazosentan | Placebo
All-Cause Mortality (participants affected / at risk) | 7/207 | 3/199
Serious Adverse Events (participants affected / at risk) | 33/207 | 26/199
Other Adverse Events (participants affected / at risk) | 156/207 | 140/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clazosentan (N=207) | Placebo (N=199)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (2)
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Brain death (General disorders) | 2 (2) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningoencephalitis herpetic (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas aeruginosa meningitis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 3 (3) | 0 (0)
Incision site discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 3 (3) | 0 (0)
Brain oedema (Nervous system disorders) | 4 (4) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 4 (4) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral microinfarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral vasoconstriction (Nervous system disorders) | 13 (15) | 12 (13)
Delayed ischaemic neurological deficit (Nervous system disorders) | 0 (0) | 1 (2)
Hydrocephalus (Nervous system disorders) | 3 (3) | 3 (3)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 1 (1)
Neurological decompensation (Nervous system disorders) | 2 (4) | 0 (0)
Posthaemorrhagic hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 2 (2)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Distributive shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clazosentan (N=207) | Placebo (N=199)
Anaemia (Blood and lymphatic system disorders) | 12 (14) | 8 (8)
Constipation (Gastrointestinal disorders) | 32 (37) | 28 (34)
Nausea (Gastrointestinal disorders) | 17 (17) | 6 (6)
Vomiting (Gastrointestinal disorders) | 17 (19) | 6 (6)
Pyrexia (General disorders) | 42 (44) | 35 (38)
Pneumonia (Infections and infestations) | 13 (13) | 6 (7)
Urinary tract infection (Infections and infestations) | 25 (25) | 24 (24)
Alanine aminotransferase increased (Investigations) | 15 (16) | 14 (14)
Aspartate aminotransferase increased (Investigations) | 13 (13) | 9 (9)
Gamma-glutamyltransferase increased (Investigations) | 24 (24) | 20 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 25 (28) | 31 (37)
Hyponatraemia (Metabolism and nutrition disorders) | 33 (34) | 29 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (10)
Cerebral vasoconstriction (Nervous system disorders) | 22 (27) | 39 (56)
Headache (Nervous system disorders) | 31 (42) | 23 (24)
Intracranial pressure increased (Nervous system disorders) | 13 (13) | 5 (5)
Insomnia (Psychiatric disorders) | 14 (14) | 11 (11)
Polyuria (Renal and urinary disorders) | 7 (8) | 10 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 2 (2)
Hypertension (Vascular disorders) | 10 (10) | 26 (28)
Hypotension (Vascular disorders) | 18 (18) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by the investigators must be submitted to the sponsor for review at least 30 days prior to submission for publication or presentation at a congress. Upon review, the sponsor may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.

DOCUMENTS (3):
  • Study Protocol: Protocol (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03585270/Prot_000.pdf
  • Study Protocol: Addendum to protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT03585270/Prot_003.pdf
  • Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT03585270/SAP_001.pdf